CLINICAL TRIAL: NCT05742659
Title: Effects of Developing a Mobile-based Interactive Simulation Scheme for Assisting the Personalized Hands-on Learning of Nasogastric Tube Insertion: a Randomized Controlled Trial
Brief Title: Effects of Developing a Mobile-based Interactive Simulation Scheme for Assisting the Personalized Hands-on Learning of Nasogastric Tube Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NCKUH-B-ER-109-194
Record Dates: First submitted 2022-12-21; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2022-12

CONDITIONS: Nasogastric Tube Insertion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Other: A mobile-based interactive simulation scheme (MISS)
- control group (No Intervention)

INTERVENTIONS:
Other: A mobile-based interactive simulation scheme (MISS) — A mobile-based interactive simulation scheme (MISS) was proposed and developed to investigate its effects on facilitating hands-on learning of NG insertion in undergraduate medical students.
  Arms: experimental group

SUMMARY:
A mobile-based interactive simulation scheme (MISS) was proposed and developed to investigate its effects on facilitating hands-on learning of nasogastric tube insertion in undergraduate medical students.

ELIGIBILITY:
Inclusion Criteria:

* fifth-year undergraduate medical students
* at least 20 years old
* without any practical clinical experience

Exclusion Criteria:

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
The 10-item evaluation questionnaire on Nasogastric tube insertion knowledge | one week
  0-100. Zero is the worst, and 100 is the best.
The self-confidence scale (C-scale) | one week
  1-5. One is high uncertainty, and five is complete certainty.

SECONDARY OUTCOMES:
System Usability Scale (SUS) | one week
  1-5. One is strongly disagree, and five is strongly agree.
The NASA-TLX (Task load index) | one week
  1-5. One is strongly disagree, and five is strongly agree.
The overall learning satisfaction | one week
  1-5 each. One is strongly disagree, and five is strongly agree. The questionnaire included 20 questions, divided into 11 categories: perceived enjoyment, comparison, diagnosis report, satisfaction, intension to use, perceived usefulness, perceived ease of use, image, output quality, result demonstrability, and cognitive load.
The OSCE (Objective Structured Clinical Examination) test | one week
  0-100. Zero is the worst, and 100 is the best.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No